CLINICAL TRIAL: NCT00663962
Title: A Prospective, Randomized, Double Blinded, Placebo Controlled Pilot Study Assessing the Effect of Perioperative Pregabalin on the Incidence of Chronic Post Thoracotomy Pain Syndrome
Brief Title: Pregabalin and Post-thoracotomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Jorge Zamora, MD, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAE-139-08
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Pain
Keywords: Thoracotomy; Post-surgical; Pregabalin
MeSH Terms: conditions — Chronic Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perioperative pregabalin (Experimental): Pregabalin 150mg administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-operatively (n=3) or Pregabalin 300mg administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-operatively (n=4).
  Interventions: Drug: Pregabalin
- Placebo control (Placebo Comparator): An identical placebo administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-op. (N=8)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — PHASE 1 (N=3) Pregabalin 150mg administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-op.
  PHASE 2 (N=4) Pregabalin 300mg administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-op.
  Arms: Perioperative pregabalin
Drug: Placebo — An identical placebo administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-op (N=8)
  Arms: Placebo control

SUMMARY:
With Institutional Ethics Board approval and signed informed consent, a pilot investigation was conducted in which 15 adult patients scheduled to undergo a thoractomy were randomly assigned to receive 1) 150 mg pregabalin 1 hour preoperatively and then 7 days postoperatively (BID) or 2) 300 mg pregabalin 1 hour preoperatively and 7 days postoperatively (BID) or 3) placebo for same regimen to assess the feasibility, safety and compliance of this drug regimen on this patient population. This assessment was necessary in order to plan a future fully powered randomized controlled trial looking at the efficacy of perioperative pregabalin ifor reducing the incidence/severity of chronic post-thoracotomy pain.

DETAILED DESCRIPTION:
Chronic post thoracotomy pain syndrome (CPTPS) is a significant problem that has important effects on patients' daily activities. The severity of postoperative pain and the central sensitization associated with it are thought to play a role in the chronification of acute pain. Gabapentin has been shown to be effective in reducing acute post-surgical pain and treating CPTPS. There is conflicting data regarding its effects on the development of chronic post-surgical pain. Although pregabalin is similar to gabapentin there are only a few studies examining its use in the modification of post-surgical pain but evidence suggests that it might be effective. There are no studies examining the effect of pregabalin on the development of chronic post-surgical pain. Our hypothesis is that perioperative use of pregabalin will decrease the incidence of CPTPS. Our ultimate goal is to conduct a multi-center study assessing the effect of perioperative oral pregabalin on the development of CPTPS. Prior to this, we will carry out a prospective, randomized, placebo controlled, double-blinded pilot study to assess the feasibility, safety, and compliance associated with perioperative use of oral pregabalin in patients undergoing video assisted thoracotomy surgery (VATS) or open thoracotomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracotomy (ET) or video assisted thoracotomy (VAT);
* Understanding and provision of written informed consent;
* Age > 18 and < 75;
* ASA class I, II or III.

Exclusion Criteria:

* Inability to adhere to study protocol;
* Intolerance or known hypersensitivity to any agents to be used in the study;
* Contraindication to thoracic epidural placement in open thoracotomy patients;
* Inability to respond to the study questionnaire;
* Renal insufficiency (serum creatinine > 1.5 x upper limit of normal);
* BMI > 40;
* Confounding procedural factors which might affect validity of data;
* Surgery for tumour extending into the chest wall;
* Requirement for second thoracotomy or re-occurrence of disease after surgery;
* Potential interaction with study medications and patient's current medications;
* Current ETOH or substance abuse;
* Pre-existing chronic pain requiring chronic analgesic use;
* History of seizure disorder requiring treatment with an anti-convulsant;
* Current therapy with thiazolidinedione class oral hypoglycemic agents (e.g. Actos, Avandia, or Avandamet);
* History of congestive heart failure;
* Major psychiatric disorder;
* Insufficient safety data in a specific patient population;
* Pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Zamora, MD, Principal Investigator — Department of Anesthesiology Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: REB approval from our institution was received to enroll 15 patients, who had given written informed consent, into this pilot study. All elective ASA I - III patients aged 18 - 75 scheduled for open thoracotomy or video assisted thoracotomy (VAT) were screened for inclusion in this study.
Pre-assignment Details: Thirty-nine patients were screened between April 23 and November 27, 2008. Fifteen patients were eligible for inclusion.
Groups:
- Placebo: An identical placebo administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-op. (N=8)
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 7 | 8
Completed | 6 (1 patient excluded for somnolence and unblinded--in 300mg group) | 8
Not Completed | 1 | 0
Not completed — somnolence | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of the 7 participants randomized to the pregabalin group, 3 receieved 150mg of pregabalin while 4 recieved 300mg pregabalin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (17.6) | 55.0 (18.6) | 57.6 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure for the Final Study Will be the Incidence of CPTPS at 2 Months.
Time Frame: 2, 4, and 6 months
Reporting Status: Not Posted

2. Primary Outcome: Incidence of Chronic Post-thoracotomy Pain at 2 Months Postoperatively
Description: Incidence of post-thoracotomy pain syndrome (persistent continuous or intermittent chest pain with resting pain score > 4 on a 10 point NRS scale)
Time Frame: 2 months postoperatively
Population: pilot study--convenience
Measure: Number; unit: participants
Groups:
- Pregabalin: Pregabalin 150mg (N=3) administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-op.
  or Pregabalin 300mg (N=4)administered one hour prior to surgery and 12 hours after surgery, then continued BID until day 7 post-op.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 7 | 8
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/7 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=7) | Placebo (N=8)
somnolence (General disorders) | 1 (1) | 0 (0) — sleepiness with 300 mg pregabalin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No